CLINICAL TRIAL: NCT01201031
Title: Reduction of Nosocomial VRE Colonization and Infection by Active Surveillance and Intervention of Infection Control (no)
Brief Title: Reduction of Nosocomial Vancomycin -Resistant Enterococci (VRE) Colonization and Infection by Active Surveillance and Intervention of Infection Control
Status: Completed | Type: Observational
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Wen-Sen Lee, Infectious Disease Department
Other Study IDs: 98105
Record Dates: First submitted 2010-09-12; First posted 2010-09-14 (Estimated); Last update posted 2011-03-16 (Estimated); Status verified 2011-03

CONDITIONS: Infection
Keywords: for the active surveillance of VRE colinization and infection
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

SUMMARY:
Vancomycin -resistant enterococci(VRE) has emerged as one of the most common nosocomial pathogen of health-care associated infection since 1988. Although the new antimicrobial agents such as Tigecycline , Daptomycin, Linezolid have clinically effectiveness for the treatment of VRE, but there was not appropriate drugs for eradicating the colonization of VRE. So the active surveillance and strict contact precaution are the best methods for VRE colonization and transmission.

This is a one year study program, we select a unit as the study site. First month (January) is the prepare period. Therefore , we collect 3 months (from February to April) baseline data, then interrupted one month(May) for the health care worker's infection control education.

Then the intervention period are three months (from June to August), and the last four months(from September to December) are the analysis and evaluation period. In the baseline period, we only do the patient's active surveillance and environmental culture. In the intervention period, beside the patient's active surveillance and environmental culture, we add contact precaution as the infection control method. If patient has VRE infection, we prescribe appropriate antibiotic therapy until the culture result proved no growth of VRE.

The aim of this study is to compare and analyze these two period (baseline period and intervention period) for understanding the transmission, risk factors and carriage rate of VRE, as the important guidelines for the VRE infection control in the future.

ELIGIBILITY:
Inclusion Criteria:

* all patients admitted to RCC unit

Exclusion Criteria:

* if the patients or family refused the exam of anal swab .

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients admitted to RCC unit , and these patients received active surveillance of VRE colinization
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2010-04; Primary Completion 2010-09 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Sen Lee, Principal Investigator — Taipei Medical University WanFang Hospital
Locations (1):
- Taipei Medical University-WanFang Hospital, Taipei, Taiwan